CLINICAL TRIAL: NCT01597934
Title: A Randomized, Multicenter, Prospective Study to Compare Antiviral Efficacy and Safety of Switching to ETV Plus TDF Versus Maintaining LAM/LDT Plus ADF Combination in CHC With PVR to LAM/LDF Plus ADF Combination Rescue Therapy for YMDD Mutation
Brief Title: Antiviral Efficacy of Switching to ETV Plus TDF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Seoul St. Mary's Hospital (Other); The Catholic University of Korea (Other); Soonchunhyang University Hospital (Other); Pusan National University Hospital (Other); Kyungpook National University Hospital (Other); Hallym University Medical Center (Other); Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hoon Ahn, Associate Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI463-274
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; Partial virologic response; YMDD mutation
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; Telbivudine; adefovir dipivoxil; entecavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: (Active Comparator): Maintaining LAM/LdT+ADV combination Lamivudine 100mg / Telbivudine 600mg +Adefovir 10mg
  Interventions: Drug: Group A (Zeffix, Sebivo, Hepsera)
- Group B (Experimental): Switching to ETV plus TDF combination Entecavir 1.0mg + Tenofovir 300mg
  Interventions: Drug: Group B (Baraclude, Viread)

INTERVENTIONS:
Drug: Group A (Zeffix, Sebivo, Hepsera) — Maintaining LAM/LdT+ADV combination Lamivudine 100mg / Telbivudine 600mg +Adefovir 10mg
  Other Names: Zeffix; Sebivo; Hepsera
  Arms: Group A:
Drug: Group B (Baraclude, Viread) — Switching to ETV plus TDF combination Entecavir 1.0mg + Tenofovir 300mg
  Other Names: Baraclude; Viread
  Arms: Group B

SUMMARY:
Switching to Entecavir(ETV) plus Tenofovir Disoproxil Fumarate(TDF) combination will result in faster and greater antiviral activity and lower rates of resistance emergence over maintaining Lamivudine(LAM)/Telbivudine(LdT)+Adefovir(ADV) combination in partial responders to LAM/LdT+ADV rescue therapy.

Earlier switching to combination with the most potent regimen will be more effective to achieve virologic response(VR) and prevent further resistance emergence.

All subjects will orally take assigned drugs once daily for 48 weeks. All subjects will be assessed at baseline and every three months thereafter. Evaluations at each visit will include vital signs, physical examinations, laboratory tests, HBV DNA levels and adverse events. At baseline and every six months thereafter, serum will be assayed for HBV serology. Genotypic analysis will be performed at baseline and 48 weeks.

DETAILED DESCRIPTION:
1. As TDF has not been approved yet in Korea, current KASL practice guideline generally recommends to add ADV in LAM-resistant or LdT-resistant patients.
2. However, several local literatures reported a substantial proportion of patients treated with LAM plus ADV combination therapy showed a persistently inadequate or partial virologic response('VR') and YMDDm still maintained in spite of under rescue combination therapy.
3. Due to the unavailability of TDF in Korea, ETV plus ADV combination has being considered a better salvage therapy with non-overlapping cross-resistance profiles in pts who fail to LAM plus ADV rescue therapy and local report demonstrated that the rate of VR was significantly higher with ETV+ADV switching group than LAM+ADV continuation group in partial responder to LAM plus ADV combination rescue therapy for LAM resistance.
4. Hence, more earlier combination therapy with the most potent Nucleoside and Nucleotide analogue would be a promising salvage treatment for previous NA treatment failures but comparative prospective trials are limited.
5. Therefore, this study will investigate the greater effectiveness and safety of switching to the most potent combination versus maintaining LAM(or LdT) plus ADV and also compare the rate of VR based on the HBV DNA cut-off level at switching - more than and less than 20,000 IU/mL.

All subjects will orally take assigned drugs once daily for 48 weeks. All subjects will be assessed at baseline and every three months thereafter. Evaluations at each visit will include vital signs, physical examinations, laboratory tests, HBV DNA levels and adverse events. At baseline and every six months thereafter, serum will be assayed for HBV serology. Genotypic analysis will be performed at baseline and 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 20 years of age
2. History of HBsAg positive for more than 6 months
3. History of genotypic resistance to LAM or LdT (YMDDm)
4. Partial responder (HBV DNA ≥ 60 IU/mL) currently receiving antiviral combination rescue therapy for at least 24 weeks of treatment with LAM+ADV or LdT+ADV
5. Hepatitis B e Antigen(HBeAg)-positive and -negative
6. Compensated liver disease (Child-Pugh A)
7. Signed written informed consent after being instructed about the objective and procedure of the clinical study

Exclusion Criteria:

1. History of genotypic resistance to ADV
2. Most previous treatment of other than LAM+ADV and LdT+ADV
3. Subjects with Alanine Aminotransferase(ALT) > 10xUpper Limit of normal(ULN)
4. Co-infected with hepatitis C virus(HCV) or HIV
5. Pregnant or lactating woman
6. Subject who needs long-term administration of drugs including immunosuppressive agents, agents related to high risk in the hepatic/renal toxicity, agents influencing renal excretion
7. History of liver transplantation or planned for liver transplantation
8. Subject who was diagnosed malignant tumor and has been receiving chemotherapy
9. Subject who has HCC history or who shows potential hepatocellular carcinoma (HCC) finding such as suspicious region in the radiologic exam(abdominal US or CT) or serum Alpha Feto Protein(AFP) elevation
10. Renal Insufficiency (CLcr < 50ml/min based on Cockcroft-Gault equation considering weight, ages and serum creatinine)
11. Subject who has a liver disease other than chronic hepatitis B (e.g. hemochromatosis, Wilson's disease, alcoholic liver disease, nonalcoholic fatty liver disease, alpha 1-antitrypsin deficiency etc.)
12. Subject who has a history of hypersensitivity to study drug or its ingredients
13. Subject who is involved in other clinical trial within 60 days prior to study entry
14. Subject who the investigator deems inappropriate to participate in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieve virologic response(HBV DNA < 60 IU/mL, approximately 300 copies/mL) by real-time PCR at Week 48 | at Week 48
  To compare the proportion of subjects who achieve virologic response(HBV DNA < 60 IU/mL, approximately 300 copies/mL) in switching group(Entecavir plus Tenofovir) with that in maintaining group(Lamivudine/Telbivudine plus Adefovir) by real-time Polymerase chain reaction(PCR) at Week 48

SECONDARY OUTCOMES:
Virologic efficacy | Week 12, 24, 36, and 48
  To compare virologic response in switching group(Entecavir plus Tenofovir) with those in maintaining group (Lamivudine/Telbivudine plus Adefovir) at Week 48
serologic efficacy | Week 12, 24, 36, and 48
  To compare serologic response in switching group(Entecavir plus Tenofovir) with those in maintaining group (Lamivudine/Telbivudine plus Adefovir) at Week 48
biochemical efficacy | Week 12, 24, 36, and 48
  To compare biochemical response in switching group(Entecavir plus Tenofovir) with those in maintaining group (Lamivudine/Telbivudine plus Adefovir) at Week 48
Safety issue | Week 12, 24, 36, and 48
  To compare safety issue in switching group(Entecavir plus Tenofovir) with those in maintaining group (Lamivudine/Telbivudine plus Adefovir) at Week 48 - severity of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Ahn, MD, PhD, Principal Investigator — Yonsei University

REFERENCES:
- [Derived] Woo HY, Park JY, Bae SH, Kim CW, Jang JY, Tak WY, Kim DJ, Kim IH, Heo J, Ahn SH. Entecavir+tenofovir vs. lamivudine/telbivudine+adefovir in chronic hepatitis B patients with prior suboptimal response. Clin Mol Hepatol. 2020 Jul;26(3):352-363. doi: 10.3350/cmh.2019.0044n. Epub 2020 May 28. PMID 32460460